CLINICAL TRIAL: NCT04514003
Title: The Corona and COVID-19 Study in Telemark and Agder - COVITA
Brief Title: The Corona and COVID-19 Study in Telemark and Agder
Acronym: COVITA
Status: Active, not recruiting | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Sorlandet Hospital HF (Other Government); Norwegian Institute of Public Health (Other Government); London School of Hygiene and Tropical Medicine (Other); Leiden University (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Anne Kristin M. Fell, Associate Professor, senior physician, Sykehuset Telemark
Other Study IDs: COVITA
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Covid19
Keywords: Immunity; Risk factors; Test-negative design; Population controls
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for SARS-CoV-2 IgG antibody testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV-2 PCR positive cases: Antibody tests will be performed every 6 months for 2 years
- SARS-CoV-2 PCR negative cases: Antibody tests will be performed at baseline
- Population controls: A large sample (n= 22500) from the general population will be included to assess risk factors. No blood sample will be collected for this group and the data needed is already collected.

SUMMARY:
Through SARS-CoV-2 IgG testing of PCR positive and negative cases the study will follow the COVID-19 immune response by monitoring the SARS-CoV-2 IgG antibody levels over a period of two years. Further, risk factors will be identified by the use of the test-negative design including population controls, allowing comparison of participants with positive and negative tests, and with population controls (triangulation). Special emphasis will be on high risk groups in general and on different occupational, environmental and socio-economic groups in particular. Finally, severity of illness, deaths and the use of health care during will be assessed using national register data from Telemark and Agder.

DETAILED DESCRIPTION:
Objectives

The main objectives are:

1. Monitor the incidence of COVID-19 and the development of the SARS-CoV-2-IgG levels of cases in Agder and Telemark over a period of two years (WP1).
2. Identify risk factors for COVID-19 by comparison of SARS-CoV-2 antibody positive and negative cases in Telemark and Agder, and comparison of these groups separately with population controls (WP2).
3. The incidence of neurocognitive symptoms and fatigue in COVID-19 patients (WP3).
4. Investigation of severity, death and the use of health care for the COVID-19 patients based on data from national registers (WP4).

The main exposures are (WP1-3):

* Infection (mild, severe) with COVID-19.
* Occupational risk factors assessed by occupational codes (ISCO88) and job exposure matrix categorisation.
* Environmental risk factors (road traffic outside bedroom window, travel by foot or bicycle alongside busy roads, and the use of a fireplaces in residential homes. Further, estimated measurements of air pollution may be linked to participants' home address.
* Socioeconomic status; age, sex, comorbidity, medication use, lifestyle factors (smoking, BMI, physical activity, others), geographic region/municipality, education and income.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years
* Performed SARS-CoV-2 PCR test

Exclusion Criteria:

* Non-Norwegian speakers.
* Deceased
* inability to answer questionnaire due to dementia or similar conditions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inhabitants of Agder and Telemark County in Norway fulfilling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 IgG antibody level | 2020-2023
  Serum Levels of SARS-CoV-2 IgG antibody and the Development of these over a two years period
Risk factors for COVID-19 | 2020-2026
  Different risk factors (age, sex, education, comorbidity, occupational and environmental exposure will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kristin M. Fell, PhD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Telemark Hospital, Skien, Vestfold and Telemark, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarjomaa M, Berg KK, Jaioun K, Tveten Y, Kersten H, Reiso H, Eikeland R, Thilesen C, Nordbo SA, Aaberge IS, Pearce N, Fell AKM. SARS-CoV-2-specific humoral immunity in a Norwegian cohort between 2020 and 2023. BMC Med. 2025 Jun 3;23(1):332. doi: 10.1186/s12916-025-04171-2. PMID 40462062